CLINICAL TRIAL: NCT03825497
Title: WALK-Copenhagen (WALK-Cph): Promoting Physical Activity in Older Adults During Hospitalization and After Discharge
Brief Title: The WALK-Copenhagen Trial (WALK-Cph): a Mixed Methods Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of inclusion
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Velux Fonden (Other); Danske Fysioterapeuter (Other)
Responsible Party: Principal Investigator, Mette Merete Pedersen, Postdoctoral Fellow, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-18027877
Record Dates: First submitted 2018-10-05; First posted 2019-01-31 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Hospitalization; Activity
Keywords: older medical patient; mobility; hospitalization; activity monitoring; cross sectoral
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A feasibility study at Medical Wards (intervention wards) in Oct 2018, January 2019 and February 2019 prior to a cluster randomized trial. Medical wards at 4 different hospitals representing clusters - 2 intervention clusters and 2 control clusters.
Masking Description: All patients at the intervention wards will receive the intervention why neither investigators nor outcome assessors will be blinded to the intervention. Patients at intervention and control wards will get equal information regarding the study and will be asked to participate in equal assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 1) On admission, patients will receive a welcome folder focusing on physical activity; 2) daily during hospitalization, patients will be encouraged to walk along a walk path in the hallway; 3) during hospitalization, patients will be encouraged to consult and use posters with exercises (sit to stand, heel raise, balance); 4) on admission, patients will receive a prescribed walk plan with 3 daily walking sessions to perform during hospitalization (3 times 1 minute, 5 minutes or 10 minutes); 5) during hospitalization patients will be motivated to pick up of clothes and beverages themselves; 6) patients will be discharged with a walk plan to use at home; 7) after discharge the municipality will follow up on patients receiving home care and patients with a rehabilitation plan
  Interventions: Other: Promotion of activity during and after hospitalization
- Usual care (No Intervention): All patients admitted to the control wards will receive usual care during and after hospitalization.

INTERVENTIONS:
Other: Promotion of activity during and after hospitalization — 1) a welcome folder encouraging physical activity; 2) encouragement to use a walk path established in the ward; 3) encouragement to use posters containing exercise suggestions;4) prescription of a walk-plan for in-hospital use; 5) encouragement to pick up clothes and beverages by oneself; 6) prescription of a walk-plan at discharge for at home use 7) follow-up on walk plan after discharge by municipality
  Arms: Intervention

SUMMARY:
The WALK-Copenhagen project aims at enhancing physical activity during and after hospitalization in older medical patients by an intervention developed in co-operation with key stakeholders

DETAILED DESCRIPTION:
In four phases we will develop (Phase 1), fidelity- and feasibility test (Phase 2), efficacy test (Phase 3) and adoption test the intervention (Phase 4). The project will use a combination of qualitative (Phase 1-4) and quantitative methods (Phase 2-3) and consists of two parallel tracks - WALK-Intervention and WALK-Implementation. Phase 1 of the study has been completed. Through workshops with patients, relatives, health professionals and researchers we have developped an intervention to enhance physical activity. Phase 2 will be carried out in October 2018 and January 2019 at Copenhagen University Hospital Hvidovre and in February 2019 at Copenhagen University Hospital, Frederiksberg. The developed intervention will be fidelity tested through daily observations at the wards. Also, the intervention will be feasibility tested in a prospective cohort study aiming at qualifying the intervention, testing recruitment strategies, testing patient willingness towards the intervention, testing randomization and blinding procedures and estimating an inclusion rate for Phase 3 (randomized controlled trial) to be conducted in 2019.

Update March 2019:

Due to a political decision to close down the medical ward at Copenhagen University Hospital, Frederiksberg in the spring of 2019, it was decided to change Phase 3 to a cohort study at Copenhagen University Hospital, Hvidovre. This decision was based on the fact that the methodological setup of the study (cluster RCT) was unintentionally changed due to the close down of one of the intervention wards.

Update November 2019:

Due to changes in characteristics of patients admitted to the intervention ward and thus a very slow inclusion rate in Phase 3 (Cohort Study), it was decided to terminate inclusion of patients. Qualitative data will still be collected as anticipated.

ELIGIBILITY:
Inclusion Criteria:

* +65 years
* acutely admitted to intervention wards
* able to walk independently with or without walking aid

Exclusion Criteria:

* in isolation
* inability to cooperate
* not able to speak or understand Danish
* in treatment for cancer
* terminally ill
* transferred to intensive care unit or another ward within 24 hours after admission

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Upright time measured by an ActivPal (PAL Technologies Ltd) activity monitor | Mean number of hours per day spent upright during hospitalization (up to 7 days)
  Between group difference in time spent standing or walking per day (Upright time)

SECONDARY OUTCOMES:
Number of steps measured by an ActivPal (PAL Technologies Ltd) activity monitor | Mean number of steps per day during hospitalization (up to 7 days)
  Between group difference in number of steps per day
Time spent lying/sitting measured by an ActivPal (PAL Technologies Ltd) activity monitor | Mean number of hours per day spent lying/sitting during hospitalization (up to 7 days)
  Between group difference time spent lying/sitting per day
Change in upright time measured by an ActivPal (PAL Technologies Ltd) activity monitor | Change in mean number of hours per day spent upright between hospitalization and 4 weeks after discharge
  Between group difference in change in time spent standing or walking per day (Upright time)
Change in number of steps measured by an ActivPal (PAL Technologies Ltd)activity monitor | Change in mean number of steps per day between hospitalization and 4 weeks after discharge
  between group difference in change in number of steps per day
Change in time spent lying/sitting measured by an ActivPal (PAL Technologies Ltd) activity monitor | Change in mean number of hours per day spent lying/sitting between hospitalization and 4 weeks after discharge
  Between group difference in change in time spent lying/sitting per day
Change in Life-Space mobility using The University of Alabama at Birmingham (UAB) Life Space Assessment (a 0-120 point scale with 0 representing low mobility and 120 high mobility) | Change in Life Space between admission and 4 weeks after discharge
  Between group difference in change in Life Space
Change in 4-meter gait speed test | Change in habitual gait speed between admission and 4 weeks after discharge
  Between group in change in Habitual gait speed
Change in mobility using The de Morton Mobility Index (DEMMI) (0-100 point scale with 0 representing low mobility and 100 representing high mobility) | Change in DEMMI score between admission and 4 weeks after discharge
  Between group difference in change in mobility

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Pedersen, PhD, Principal Investigator — Postdoc, Clinical Research Centre, Hvidovre Hospital, Denmark
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Derived] Pedersen BS, Kirk JW, Olesen MK, Gronfeldt BM, Stefansdottir NT, Brodsgaard R, Tjornhoj-Thomsen T, Nilsen P, Andersen O, Bandholm T, Pedersen MM. Feasibility and implementation fidelity of a co-designed intervention to promote in-hospital mobility among older medical patients-the WALK-Copenhagen project (WALK-Cph). Pilot Feasibility Stud. 2022 Apr 9;8(1):80. doi: 10.1186/s40814-022-01033-z. PMID 35397574
- See also: A tailored strategy for designing the Walk-Copenhagen (WALK-Cph) intervention to increase mobility in hospitalised older medical patients: a protocol for the qualitative part of the WALK-Cph project — https://bmjopen.bmj.com/content/8/3/e020272